CLINICAL TRIAL: NCT06238804
Title: Characteristic Analysis and Surgical Exploration for Acetabular Roof Fractures: Multicenter Retrospective Cohort Study
Acronym: CASEARF
Status: Withdrawn | Type: Observational
Why Stopped: Due to limited funding, the study is now being withdrawn.
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Principal Investigator, Ruipeng Zhang, Doctor, Hebei Medical University Third Hospital
Other Study IDs: ZRP2024
Record Dates: First submitted 2024-01-23; First posted 2024-02-02 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fracture types: A3.1, A3.2, A3.3
  Interventions: Procedure: KL, Iliofemoral, Ilioinguinal, Iliac fossa and combined approaches

INTERVENTIONS:
Procedure: KL, Iliofemoral, Ilioinguinal, Iliac fossa and combined approaches — A3.1, A3.2, A3.3
  Other Names: Fracture types

SUMMARY:
Acetabular roof was a crucial structure for maintaining the stability of hip joint; however, its important role was not especially emphasized in the Letournel-Judet classification system. Acetabular roof was segmented into the roof column and roof wall in Three-column classification and fracture in this area alone was defined as A3 injury. Radiographic data and functional outcome of A3 injury patients were reviewed to explore the characteristics and surgical strategy.

DETAILED DESCRIPTION:
Fracture data, surgical incision, operation time, blood loss, fracture healing， Reduction quality，functional outcome，and relevant complications

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years, acute (<14 days) closed roof column/wall acetabular fractures (A3.1, A3.2 or A3.3) in Three-column classification, normal activity of the affected hip before the injury, received surgical reduction and internal fixation

Exclusion Criteria:

* open fractures, pathologic fractures, limited range of motion (ROM) of the hip joint before the injury, conservative treatment, risk factors affecting bone healing (such as smoking and metabolic diseases) and noncompletion of the two-year follow-up

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients met the inclusion criteria were collected in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
postoperative outcome | 4 months
  Merle d'Aubigné score, fracture healing, reduction quality, etc

SECONDARY OUTCOMES:
complication | 1 month
  wound infection, iatrogenic injury of vessels and nerves, etc

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Hou, MD, Study Chair — Hebei Medical University Third Hospital
Locations (1):
- Hebei Medical University Third Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No
The datasets used and analyzed during the current study are available from the corresponding author on reasonable request.